CLINICAL TRIAL: NCT02492503
Title: An Open Label Randomized Phase 2, Pilot Study to Investigate the Effectiveness of Palliative Chemotherapy in Stage IVB, Recurrent or Persistent Carcinoma Cervix
Brief Title: Effectiveness of Chemotherapy in Metastatic or Recurrent Carcinoma Cervix
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Harish P, senior resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA CX CHEMOTHERAPY
Record Dates: First submitted 2014-01-08; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Metastatic Carcinoma to the Uterine Cervix; Recurrent Carcinoma Cervix; Cervix Carcinoma Recurrent
Keywords: recurrent or metastatic carcinoma cervix chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence | interventions — Paclitaxel; Carboplatin; 26S proteasome non-ATPase regulatory subunit 13; DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pacli carb 3 (Active Comparator): Paclitaxel 175 mg/ m2 administered in 250 ml normal saline over 3 hours and carboplatin AUC 4-5 administered in 250 ml 5%D over 2 hours. Therapy repeated every three weekly
  Interventions: Drug: Paclitaxel and carboplatin
- pacli carb 1 (Active Comparator): Paclitaxel 60 mg/ m2 administered in 250 ml normal saline over 1 hour and carboplatin AUC 2 administered in 250 ml 5%D over 1 hour. Therapy repeated every weekly
  Interventions: Drug: Paclitaxel and carboplatin

INTERVENTIONS:
Drug: Paclitaxel and carboplatin — Paclitaxel 60 mg/ m2 administered in 250 ml normal saline over 1 hour, and carboplatin AUC 2 administered in 250 ml 5%D over 1 hour. Therapy repeated every weekly
  Other Names: Arm1
  Arms: pacli carb 1
Drug: Paclitaxel and carboplatin — Paclitaxel 175 mg/ m2 administered in 250 ml normal saline over 3 hours and carboplatin AUC 4-5 administered in 250 ml 5%D over 2 hours. Therapy repeated every three weekly
  Other Names: Arm 2
  Arms: pacli carb 3

SUMMARY:
Experience with substituting carboplatin for cisplatin is limited in advanced and recurrent cervix cancer and there has been no counterpart to GOG 158, which documented therapeutic equivalency of cisplatin/paclitaxel and carboplatin/paclitaxel for treatment of ovarian cancer, performed in a cervix cancer population.

DETAILED DESCRIPTION:
This trial will be a prospective, randomized phase II pilot study. Consecutive patients of metastatic, recurrent or refractory carcinoma cervix enrolled in gynecology clinic at IRCH, AIIMS will be taken into study after taking informed consent. Patients will be randomized into two arms. Each arm shall contain 20 patients. The patients shall receive paclitaxel and carboplatin q3wk in first arm and paclitaxel and carboplatin q1 wk in second arm.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven case of squamous or adenocarcinoma or adenosquamous carcinoma 2.ECOG performance status 0,1 and 2 3.Adequate hematologic, renal and liver functions 4.Informed consent 5.Measurable disease by CT scan or USG abdomen or MRI

-

Exclusion Criteria:

1. ECOG performance status 3 or 4
2. Impaired blood counts: those patients with an absolute neutrophil count <1,500/μL, platelet counts <100,000/μL, will be ineligible.
3. Impaired renal /liver functions as indicated by:

Serum bilirubin >1.5× normal, AST level more than 3× normal, Alkaline phosphatase level more than 3× institutional normal, or a Serum creatinine level more than 1.2 mg/dL. Patients with serum creatinine level of more than 1.2 mg/dL but less than 1.5 mg/dL are eligible if creatinine clearance is 70 ml/min were eligible if a creatinine clearance determination was more than 50 mL/min.

4. H/o prior chemotherapy for metastatic disease, 5. H/O concurrent or past malignancy other than carcinoma cervix, 6. CNS metastasis, or 7. Bilateral hydronephrosis that could not be alleviated by ureteral stents or percutaneous nephrostomy.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Time to progression (length of time from start of chemotherapy to evidence of cancer progression. | 6 months

SECONDARY OUTCOMES:
Response rate | 6 months
Overall survival | 6 months
Quality Of Life Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: lalit kumar, MD,DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, New Delhi, India

REFERENCES:
- See also: Witteveen PO et al — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2731017/